CLINICAL TRIAL: NCT04116372
Title: Increasing Physical Activity in Empty Nest and Retirement Populations: A Feasibility Trial of an Online Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Victoria (Other)
Responsible Party: Principal Investigator, Ryan Rhodes, Professor Ryan Rhodes, University of Victoria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 05-281982
Record Dates: First submitted 2019-10-03; First posted 2019-10-04 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Physical Activity; Health Promotion
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Empty Nest Intervention Group (Experimental): Participants will complete a baseline questionnaire, and receive access to the our online platform for 10 weeks. Completing the online platform is designed to encourage participants to engage in physical activity. At 2 and 5 weeks, a check-in session will occur over the phone. At 10 weeks the participant will be contacted to return to the lab to complete the final questionnaire, and do a wrap up interview. The end-of-trial qualitative interview will evaluate participant satisfaction and feasibility of the intervention. For this reason a lab employee unaffiliated with this study will complete these in person interviews.
  Interventions: Behavioral: Digital Health Online Platform
- Retirement Intervention Group (Experimental): Participants will complete a baseline questionnaire, and receive access to the our online platform for 10 weeks. Completing the online platform is designed to encourage participants to engage in physical activity. At 2 and 5 weeks, a check-in session will occur over the phone. At 10 weeks the participant will be contacted to return to the lab to complete the final questionnaire, and do a wrap up interview. The end-of-trial qualitative interview will evaluate participant satisfaction and feasibility of the intervention. For this reason a lab employee unaffiliated with this study will complete these in person interviews.
  Interventions: Behavioral: Digital Health Online Platform
- Empty Nest Control Group (No Intervention): This group will complete baseline and final questionnaires (online or paper). At the end of the study this group will have the option to receive access to the other group's materials (online platform) if they wish, for the 10 week period following the study.
- Retirement Control Group (No Intervention): This group will complete baseline and final questionnaires (online or paper). At the end of the study this group will have the option to receive access to the other group's materials (online platform) if they wish, for the 10 week period following the study.

INTERVENTIONS:
Behavioral: Digital Health Online Platform — The website has 10 lessons that the participant will gain access to on a weekly basis. Lesson titles are as follows:
  Lesson 1 - Benefits of Physical Activity on Chronic Disease Lesson 2 - Mental benefits of Physical Activities Lesson 3 - Increasing Self Confidence for Physical Activities Lesson 4 - Learning about your Emotions Lesson 5 - Building Social Support Lesson 6 - Building Physical Activity Opportunity Lesson 7 - Goal Setting and Planning Lesson 8 - Self Monitoring Lesson 9 - Habit Lesson 10 - Identity
  Arms: Empty Nest Intervention Group; Retirement Intervention Group

SUMMARY:
Internet-based health promotion programs have the potential to reach more individuals than in person interventions, without overtaxing healthcare resources. Having a high quality, user-centered web-based program can help maximize user engagement and adherence. Thus, the primary objective of this pilot study is to examine the feasibility and acceptability of a web-based physical activity behavior change program on recently retired and/or empty nest populations. The primary research question is: Is it worthwhile to conduct a larger scale eHealth study targeting empty nest and/or retired populations based on preliminary results and feedback from this pilot study. We will also be examining changes other behavioral indicators related to physical activity as a secondary outcome measure.

DETAILED DESCRIPTION:
Background: Physical activity is associated with management and/or prevention of over 25 chronic health conditions; however the majority of adults in North America are not active enough to experience these benefits. Behavioral strategies have been shown to be effective for increasing physical activity, and our online platform includes components of several behavioral strategies including goal setting and feedback.

Target Population: Sedentary adults who have recently (within 6 months of enrollment) retired, or had their last child leave the family home, living in Victoria, British-Columbia, Canada.

Sample Size: 80 participants, 20 participants per group - Empty Nest (Control) Empty Nest (intervention), Retired (Control), Retired (Intervention).

Intervention: Participants in each Empty Nest and Retirement participant pool will be randomized to two groups: 1 - Waitlist control group, 2 - Access to Online Platform. Half of the empty nest participant group and half of the retired participant group will receive an intervention, with the other half representing the control comparison group. Participants from both groups will complete an online questionnaires at baseline and 10 weeks. The intervention group will also be asked for an in-person exit interview.

ELIGIBILITY:
Inclusion Criteria:

Potential participants will be included if they have either a) recently (within 6 months) retired, or b) experienced children moving out of the familial home. In addition, potential participants must have access to the internet at home, and have a smart phone or home computer that can support the eHealth application we are using. Potential participants must currently be not meeting the physical activity (PA) guidelines (less than 150 minutes of moderate to vigorous aerobic activity). There will be no delimitations to the sample based on socio-economic or ethnic variables.

Exclusion Criteria:

Participants will be excluded from the project if they not have access to the Internet, are unable to speak/read English, are engaging in moderate-to vigorous PA (MVPA) sufficient to meet the PA Guidelines, have an existing chronic medical condition potentially making them at risk of injury or ill health from increasing their physical activity (assessed using the GAQ)

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Recruitment rate (monthly) | 4 months
  For the full scale RCT, we are looking for a 1 day per week or 30 min MVPA change which equates to an approximate effect size of d = .35. This equates to roughly 65 per group (130 for a two group trial). If we recruit for 2 years in the large trial (assuming a six month time period for each person in the intervention) we need to be recruiting at least 6 per month. If we decide on a three armed trial, we will need to recruit at least 8 per month.
Participant retention | 10 weeks
  Number of participants who complete both baseline and end of study (10 week) measures. A 80-100% retention rate is indicative of a strong trial (Jackson & Waters, 2005).
Participant intervention satisfaction/evaluation | 10 weeks
  For satisfaction ratings, mean and standard deviations will be calculated for the quantitative satisfaction and evaluation questionnaire. Given that scores of 1 (ex. not helpful, did not use the tools) and 2 (ex. Somewhat helpful, used a little bit of the tools) indicated levels of dissatisfaction, and 3 (ex. Quite helpful, used a bit of the tools) and 4 (ex. Extremely helpful, used a lot of the tools) indicated some sort of satisfaction, a mean score of ≥ 2.5 will be deemed acceptable for recommendation for a full RCT.

SECONDARY OUTCOMES:
Change in self-reported physical activity from baseline to 10 weeks | Baseline - 10 weeks
  Measured from questionnaire using Godin's personal self report leisure time measurement tool, also known as the Leisure Score Index (LSI). The Leisure Score Index contains three questions, which assess the frequency of mild, moderate, and strenuous activity performed for at least 10 minutes during free time in a typical week. Changes in these measures will be examined
Change in physical activity beliefs, attitudes, barriers, and motivation from baseline to 10 weeks. | Baseline - 10 weeks
  Included in questionnaire - Ajzen's theory of planned behaviour questionnaire will be applied to measure participants' beliefs, attitudes, barriers, and motivation related to physical activity.
Change in physical activity behaviour regulation from baseline to 10 weeks. | Baseline - 10 weeks
  Included in questionnaire - 5 items adapted from Umstattd's scale measuring physical activity self-regulation strategies in older adults. Changes in this measure will be examined
Change in physical activity habits from baseline to 10 weeks. | Baseline - 10 weeks
  Included in questionnaire - 12 Self Report Habit Index items from the measure developed by Verplanken and Orbell and adapted to physical activity by Chatzisarantis and Hagger. Changes in this measure will be examined
Change in physical activity identity from baseline to 10 weeks. | Baseline - 10 weeks
  Included in questionnaire - Anderson and Cychosz Exercise Identity Scale is used to measure participants' identification as someone who participates in physical activity.
Change in quality of life measured using the Short Form 12 questionnaire. | Baseline - 10 weeks
  The online questionnaire will asses participants' quality of life using the short form 12 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- UVIC, Victoria, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jackson N, Waters E; Guidelines for Systematic Reviews in Health Promotion and Public Health Taskforce. Criteria for the systematic review of health promotion and public health interventions. Health Promot Int. 2005 Dec;20(4):367-74. doi: 10.1093/heapro/dai022. Epub 2005 Sep 16. PMID 16169885